CLINICAL TRIAL: NCT01642485
Title: Evaluation of the Effect of Different Foods, Carbohydrate Meal, and a Euglycaemic Insulin Clamp on the QT/QTc Interval Using a Single Dose of Moxifloxacin as a Positive Control in Healthy Male and Female, Caucasian and Japanese Volunteers
Brief Title: Food and Insulin Effect on QT/QTC Interval of ECG
Acronym: C11035
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RPL-01-11; 2011-002423-17 (EudraCT Number)
Record Dates: First submitted 2012-06-19; First posted 2012-07-17 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Effects of Different Meals on the QT/QTc Interval; Insulin and Oral Hypoglycemic [Antidiabetic] Drugs Causing Adverse Effects in Therapeutic Use; C-Peptide Effects on the QT/QTc Interval; Moxifloxacin ECG Profile in Fed and Fasted State; Japanese vs. Caucasian TQT Comparison
Keywords: Insulin clamp; Glucose clamp; Moxifloxacin; Fed; Fasted; QT/QTC interval; TQT; ECG; Meal effects; C Peptide; Japanese Caucasian bridging; TQT bridging; FDA standard breakfast; Adaptive study design
MeSH Terms: conditions — Insulin Resistance; Fasting; Lecithin Cholesterol Acyltransferase Deficiency | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin 400 mg fasted (Active Comparator): Moxifloxacin 400 mg fasted was administered on Day 3. For Day 1 and 2, there were 4 different sequences: Placebo and Insulin Clamp; Insulin Clamp and Continental breakfast; Continental breakfast and FDA breakfast; FDA breakfast and Placebo. Additionally, Caucasian vs Japanese subjects were analysed.
  Interventions: Drug: Moxifloxacin 400 mg fasted; Other: FDA breakfast; Other: Continental breakfast; Procedure: Insulin Clamp; Drug: Placebo
- Moxifloxacin 400 mg fed (Experimental): Moxifloxacin 400 mg fed was administered on Day 3 after Continental breakfast. For Day 1 and 2, there were 4 different sequences: Placebo and Insulin Clamp; Insulin Clamp and Continental breakfast; Continental breakfast and FDA breakfast; FDA breakfast and Placebo.
  Additionally, Caucasian vs Japanese subjects were analysed.
  Interventions: Other: FDA breakfast; Other: Continental breakfast; Drug: Moxifloxacin 400 mg fed; Procedure: Insulin Clamp; Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin 400 mg fasted — Subjects receiving drug (400 mg moxifloxacin),having fasted overnight for 10 hours.
  This is the standard probe for the assessment of assay sensitivity in Thorough QT (TQT) studies.
  Other Names: Moxifloxacin
  Arms: Moxifloxacin 400 mg fasted
Other: FDA breakfast — Calorie reduced FDA standard breakfast (58% fat, low carbohydrates)- On the assumption that increases in C-peptide levels are responsible for the QTc shortening observed after a meal, a lesser effect on QTc compared to a carbohydrate rich breakfast should be observed.
Other: Continental breakfast — High carbohydrate breakfast (>70% carbohydrates)- On the assumption that increases in C-peptide levels are responsible for the QTc shortening observed after a meal, a greater effect on QTc compared to a low carbohydrate breakfast (FDA standard breakfast) should be observed.
Drug: Moxifloxacin 400 mg fed — Currently, there is no published data showing the effects of a single 400 mg oral dose of moxifloxacin on the ECG/QT/QTc after food.
  Other Names: Moxifloxacin
  Arms: Moxifloxacin 400 mg fed
Procedure: Insulin Clamp — A euglycaemic/hyperinsulinaemic clamp, (DeFronzo, 1979) involves acutely raising the plasma insulin levels to a steady state and maintaining a state of euglycaemia with a glucose infusion, thereby effectively stopping endogenous insulin and C-peptide release. This technique will confirm whether hyperinsulinaemia has any effect on the QT/QTc interval.
Drug: Placebo — Comparison of different meals effect on Moxifloxacin PK profile

SUMMARY:
Moxifloxacin is routinely used as a probe to confirm assay sensitivity in thorough electrocardiogram (ECG) studies. It has been shown that a meal shortens the QT interval, which may affect pharmacokinetics (PK) and/or pharmacodynamics (PD) of the study drug. However, there is no published data clarifying this issue. There is also a paucity of data investigating ethnic differences of the effects of medicines on QTc.

The aims of the study were to compare the effect of different food contents to placebo on the changes in ECG and to demonstrate the effect of insulin, C-peptide and glucose on the ECG. This was done by giving different treatments on separate days, which included intravenous insulin, a high carbohydrate breakfast [>70%], and a calorie reduced low carbohydrate American FDA standard breakfast. Moxifloxacin 400 mg was used as a positive control and was given with and without food to Caucasian and Japanese volunteers to investigate racial differences.

DETAILED DESCRIPTION:
This study was initially performed in 24 healthy Caucasian and Japanese volunteers with an option to increase the sample size to up to 54 volunteers. The decision to increase the sample size to 32 was based on the standard deviation of the ECG intervals observed in the first 24 volunteers. This analysis was performed by an independent statistician under blinded conditions.

Each volunteer participated in 2 periods. Each period consisted of 1 baseline day (D-1) followed by 3 study days (D1 - D3) when the various food effect and drug treatments or placebo were administered. All volunteers received all treatments. Moxifloxacin was always given on D3 to prevent any carryover effect and there was a minimum washout period of 3 days in between the 2 periods.

How well the treatments (insulin/glucose, high carbohydrate breakfast, calorie reduced breakfast and moxifloxacin) were tolerated by the volunteers was assessed and any side effects noted.

We compared the effects of the various treatments between Caucasian and Japanese volunteers.

Moxifloxacin and placebo were given to volunteers by mouth, i.e. they were asked to swallow them with water. The different types of breakfast were provided which volunteers were asked to eat. Insulin and glucose were administered intravenously (Insulin/glucose clamp). Hence, the study was performed as an open-label design.

This study was conducted as a single site study at Richmond Pharmacology/ St George's University of London.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 20 - 45 years old
2. Signed ICF
3. Japanese - a descendant of four Japanese grandparents, carrying a Japanese passport and has not been outside Japan for more than 5 years prior to screening
4. The Caucasian - light to brown skin pigmentation; straight to wavy or curly hair; indigenous to Europe, northern Africa, western Asia, and India. The study may also include Caucasians from North America, Australia and South Africa
5. No clinical findings on the physical examination
6. Body mass index (BMI) = 18 - 25 kg/m2, body weight at least 48 kg.
7. Systolic blood pressure 90-145 mmHg, diastolic blood pressure 40-90 mmHg, and heart rate 40-90 bpm
8. Triplicate 12 lead ECG without clinically relevant abnormalities
9. 24 hour 12 lead Holter ECG without clinically relevant abnormalities
10. Haematology, biochemistry and urinalysis within the normal range
11. Must agree to use acceptable methods of contraception

Exclusion Criteria:

1. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug
2. History of clinically significant syncope.
3. Family history of sudden death.
4. Family history of premature cardiovascular death.
5. Family history of congenital long QT syndrome or Brugada's syndrome.
6. History of arrhythmias and ischemic heart disease
7. Conditions predisposing to electrolyte imbalances (e.g. altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa).
8. Abnormal ECG in the standard 12-lead ECG and 24-hour 12 lead Holter ECG
9. Abnormal rhythm, conduction or morphology of resting ECG, such as:

   * Sinus node dysfunction.
   * Clinically significant PR (PQ) interval prolongation.
   * Intermittent second or third degree AV block.
   * Incomplete or complete bundle branch block.
   * Abnormal T wave morphology.
   * Prolonged QTcB >450 msec or shortened QTcB < 350 msec or family history of long QT syndrome.
10. Abnormal blood glucose result (blood glucose >7.8mmol/l)
11. Significant family history of diabetes mellitus.
12. Significantly elevated fasting blood glucose level
13. Signs and/or symptoms of acute illness in the four-week period prior to screening.
14. Veins unsuitable for intravenous puncture or cannulation on either arm
15. Known hypersensitivity to any medicines administered in the trial.
16. Treatment with any prescribed medication during the 2 weeks prior to first baseline day.
17. Treatment with any over-the-counter (OTC) medications during the 2 weeks prior to first baseline day.
18. Treatment with vitamins and/or minerals within 48 hours prior to the first baseline day.
19. Treatment with another investigational drug within 4 weeks prior to dosing or having participated in more than 3 investigational drug studies within a year prior to dosing.
20. Positive urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates and methadone) or the alcohol breath test
21. History or clinical evidence of alcoholism (regular weekly alcohol intake of more than 14 units if female and 21 units if male) or drug abuse (compulsive, repetitive and/or chronic use of drugs or other substances with or without problems related to their use and/or where stopping or a reduction in dose will lead to withdrawal symptoms)
22. Excessive caffeine consumption (≥800 mg per day)
23. Smoking within 3 months prior to screening
24. Loss of 250 mL or more blood within 3 months prior to screening.
25. Positive results from the hepatitis serology, except for vaccinated subjects.
26. Positive results from the HIV serology.
27. Any circumstances or conditions, which may affect full participation in the study or compliance with the protocol.
28. Legal incapacity or limited legal capacity.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD FRCA FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, Tooting, United Kingdom

REFERENCES:
- [Background] Taubel J, Wong AH, Naseem A, Ferber G, Camm AJ. Shortening of the QT interval after food can be used to demonstrate assay sensitivity in thorough QT studies. J Clin Pharmacol. 2012 Oct;52(10):1558-65. doi: 10.1177/0091270011419851. Epub 2011 Nov 8. PMID 22067197
- [Background] Scott EM, Greenwood JP, Vacca G, Stoker JB, Gilbey SG, Mary DA. Carbohydrate ingestion, with transient endogenous insulinaemia, produces both sympathetic activation and vasodilatation in normal humans. Clin Sci (Lond). 2002 May;102(5):523-9. PMID 11980571
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Result] Taubel J, Ferber G, Lorch U, Batchvarov V, Savelieva I, Camm AJ. Thorough QT study of the effect of oral moxifloxacin on QTc interval in the fed and fasted state in healthy Japanese and Caucasian subjects. Br J Clin Pharmacol. 2014 Jan;77(1):170-9. doi: 10.1111/bcp.12168. PMID 23713767
- [Result] Taubel J, Lorch U, Ferber G, Singh J, Batchvarov VN, Savelieva I, Camm AJ. Insulin at normal physiological levels does not prolong QT(c) interval in thorough QT studies performed in healthy volunteers. Br J Clin Pharmacol. 2013 Feb;75(2):392-403. doi: 10.1111/j.1365-2125.2012.04376.x. PMID 22775199
- See also: The FIRST to obtain MHRA Standard and Supplementary Accreditation for two hospital based clinical trial units. — http://www.richmondpharmacology.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Period1:
  Day 1: Placebo Day 2: Insulin Clamp Day 3: Moxiloxacin 400 mg fasted Washout period: 3 days
  Period 2:
  Day 1: Continental breakfast Day 2:FDA breakfast Day 3: Moxifloxacin 400 mg fed (with continental breakfast)
- Sequence 2: Period1:
  Day 1: Insulin Clamp Day 2: Continental breakfast Day 3: Moxiloxacin 400 mg fasted Washout period: 3 days
  Period 2:
  Day 1: FDA breakfast Day 2: Placebo Day 3: Moxifloxacin 400 mg fed (with continental breakfast)
- Sequence 3: Period1:
  Day 1: Continental breakfast Day 2: FDA breakfast Day 3: Moxiloxacin 400 mg fasted Washout period: 3 days
  Period 2:
  Day 1: Placebo Day 2: Insulin Clamp Day 3: Moxifloxacin 400 mg fed (with continental breakfast)
- Sequence 4: Period1:
  Day 1: FDA breakfast Day 2: Placebo Day 3: Moxiloxacin 400 mg fasted Washout period: 3 days
  Period 2:
  Day 1: Insulin Clamp Day 2: Continental breakfast Day 3: Moxifloxacin 400 mg fed (with continental breakfast)
- Sequence 5: Period1:
  Day 1: Placebo Day 2: Insulin Clamp Day 3: Moxiloxacin 400 mg fed (with continental breakfast) Washout period: 3 days
  Period 2:
  Day 1: Continental breakfast Day 2:FDA breakfast Day 3: Moxifloxacin 400 mg fasted
- Sequence 6: Period1:
  Day 1: Insulin Clamp Day 2: Continental breakfast Day 3: Moxiloxacin 400 mg fed (with continental breakfast) Washout period: 3 days
  Period 2:
  Day 1: FDA breakfast Day 2: Placebo Day 3: Moxifloxacin 400 mg fasted
- Sequence 7: Period1:
  Day 1: Continental breakfast Day 2: FDA breakfast Day 3: Moxiloxacin 400 mg fed (with continental breakfast) Washout period: 3 days
  Period 2:
  Day 1: Placebo Day 2: Insulin Clamp Day 3: Moxifloxacin 400 mg fasted
- Sequence 8: Period1:
  Day 1: FDA breakfast Day 2: Placebo Day 3: Moxiloxacin 400 mg fed (with continental breakfast) Washout period: 3 days
  Period 2:
  Day 1: Insulin Clamp Day 2: Continental breakfast Day 3: Moxifloxacin 400 mg fasted
Period: Period 1, Day 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 4 (crossover so all subjects had this treatment) | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 1, Day 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 1, Day 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Day 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Day 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Day 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study population consisted of healthy non-smoking, subjects. Electrocardiograms in the placebo arm were recorded twice in fasted and fed condition.
Groups:
- All Study Participants: Subjects participating in the study attended for screening, two treatment periods (periods 1 and 2) of 4 assessment days each and a follow-up visit. Data obtained on study days 1 and 2 compared the ECG effects of different types of food and placebo. Each period consisted of a baseline ECG day (day -1) and treatment days (days 1-3). Moxifloxacin was given in fasted condition or with Continental breakfast, on day 3 of each study period. The two periods were separated by at least 3 days to allow for the effects of moxifloxacin to wash-out. No wash-out was required between the other treatments investigated. The ECG and samples for PK and PD analysis on the treatment days were taken at the corresponding clock time points as on the baseline days. Each subject received all treatments and all the comparisons between treatment effects were made intra-individually reducing the anticipated variability and thereby reducing the sample size.
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years]
  Caucasian | 25.6 (4.7)
  Japanese | 27.6 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13
  Japanese | 19
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32
Body Mass Index [Number; unit: participants]
  >18 kg/m^2 | 32
  >25 kg/m^2 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Food (Fasted and Fed State) on the Degree of QT Prolongation Caused by Moxifloxacin
Description: The primary baseline corrections were calculated using averaged QTc baseline values (the mean of all median readings recorded for each time-point on the baseline Day -1). This single value (QTcbaselineAV) was used to calculate ΔQTc for each study period.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4 and 6 hours post-dose
Population: Since the baseline was used as a covariate in the analysis, using the standard deviation of the change from baseline, in the simple sample size formula is justified. Assuming a standard deviation of 7 msec for the single differences, sample sizes for the sum can therefore work with a standard deviation of 6.5 msec.
Measure: Mean (90% Confidence Interval); unit: ms
Groups:
- Fasted Group: This study was designed as an open-label, randomized, placebo-controlled, crossover trial that evaluated the effect of a 400 mg oral dose of moxifloxacin in fasted conditions to a baseline and a placebo treatment. Data obtained on study days 1 and 2 compared the ECG effects of different types of food and placebo. Each period consisted of a baseline ECG day (day -1) and treatment days (days 1-3). Moxifloxacin was given in either the fed or fasted condition, on day 3 of each study period. The two periods were separated by at least 3 days to allow for the effects of moxifloxacin to wash-out. The ECG and samples for PK and PD analysis on the treatment days were taken at the corresponding clock time points as on the baseline days. Each subject received all treatments and all the comparisons between treatment effects were made intra-individually reducing the anticipated variability and thereby reducing the sample size.
- Fed Group: This study was designed as an open-label, randomized, placebo-controlled, crossover trial that evaluated the effect of a 400 mg oral dose of moxifloxacin in fed conditions to a baseline and a placebo treatment. Data obtained on study days 1 and 2 compared the ECG effects of different types of food and placebo. Each period consisted of a baseline ECG day (day -1) and treatment days (days 1-3). Moxifloxacin was given in either the fed or fasted condition, on day 3 of each study period. The two periods were separated by at least 3 days to allow for the effects of moxifloxacin to wash-out. The ECG and samples for PK and PD analysis on the treatment days were taken at the corresponding clock time points as on the baseline days. Each subject received all treatments and all the comparisons between treatment effects were made intra-individually reducing the anticipated variability and thereby reducing the sample size.
Arm/Group | Fasted Group | Fed Group
Number analyzed (Participants) | 32 | 32
ms | 14.4 [11.9 to 16.8] | 11.6 [9.1 to 14.1]
Statistical Analysis 1: Comparison: Fasted Group; The effect of insulin, C-peptide and glucose on QTcF was investigated using linear mixed effect concentration-response models with the double difference of QTcF (difference to time matched placebo of the change from average baseline) as dependent variable and up to two of the variables change from time matched placebo in insulin, C-peptide and glucose as covariates; Test type: Superiority or Other; p = 0.05, t-test, 1 sided

2. Secondary Outcome: The Food Effects (Calorie Reduced FDA Breakfast and Carbohydrate Rich Continental Style) on QTcF
Description: Scott et al (2002) demonstrated an increase in the heart rate of 10bpm in some healthy subjects following ingestion of a carbohydrate meal. There was significant correlation between the resultant hyperinsulinaemia and an increase in skeletal muscle blood flow, and sympathetic activity, with a reduction in vascular resistance.
  If postprandial insulinaemia is a significant influence on the QT interval, then carbohydrate rich meals would be expected to show greater effect. Therefore, to explore this on two separate days of the study subjects will be given one of two different types of breakfast:
  1. A high carbohydrate content breakfast, (>70% carbohydrate)
  2. A reduced calorie FDA standard breakfast, (58% fat, low carbohydrate content) to determine effect on QT interval.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4 and 6 hours post-dose
Measure: Mean (90% Confidence Interval); unit: ms
Groups:
- Continental Breakfast: Continental breakfast: High carbohydrate breakfast (>70% carbohydrates)- On the assumption that increases in C-peptide levels are responsible for the QTc shortening observed after a meal, a greater effect on QTc compared to a low carbohydrate breakfast (FDA standard breakfast) should be observed.
  QTcF change from a baseline presented.
- Placebo at Baseline: a baseline QTcF measured on Day -1 of each period
Arm/Group | FDA Breakfast | Continental Breakfast | Placebo at Baseline
Number analyzed (Participants) | 32 | 32 | 32
ms | -6.8 [-9.3 to -4.3] | -7.9 [-10.4 to -5.5] | 412.4 [407.9 to 416.9]
Statistical Analysis 1: Comparison: FDA Breakfast vs Continental Breakfast; The relevant confirmatory null hypotheses could all be rejected on the 5% level (one sided), i.e. a difference in QTcF between continental breakfast and placebo; between FDA breakfast and placebo could be ascertained; Test type: Superiority or Other; p = 0.05, t-test, 1 sided
Statistical Analysis 2: Comparison: Continental Breakfast; Test type: Superiority or Other; Mean Difference (Final Values) = -7.9, 90% CI 2-sided [-10.4 to -5.5]
Statistical Analysis 3: Comparison: FDA Breakfast; Test type: Superiority or Other; Median Difference (Final Values) = -6.8, 90% CI 2-sided [-9.3 to -4.3]

3. Secondary Outcome: Moxifloxacin 400 mg (Single Dose) Compared to Placebo on the Mean QT/QTc Interval.
Description: "Moxifloxacin 400mg Fasted" group is reporting the maximum change in QT/QTc interval from placebo treatment.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4 and 6 hours post-dose
Measure: Mean (90% Confidence Interval); unit: ms
Groups:
- Moxifloxacin 400 mg Fasted: The highest change was at 2.5h time point, which is presented here.
- Placebo: Time matched absolute value for QTcF for placebo treatment.
Arm/Group | Moxifloxacin 400 mg Fasted | Placebo
Number analyzed (Participants) | 32 | 32
ms | 14.4 [11.9 to 16.8] | 414.2 [409.6 to 418.8]

4. Secondary Outcome: Insulin, Glucose and C-Peptide Effects on the QT/QTc Interval
Description: The effect on QTc was investigated using linear mixed effect models with placebo corrected QTcF (change from average baseline) as a dependent variable and insulin, glucose and C-peptide (placebo corrected) as covariates for the data obtained under the euglycaemic clamp as well as for all data obtained under the clamp and the two types of breakfast.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4 and 6 hours post-dose
Measure: Median (95% Confidence Interval); unit: msec
Groups:
- Insulin Clamp; Glucose: A euglycaemic/hyperinsulinaemic clamp was used to stop any endogenous C-peptide and insulin production. The clamp acutely raised the plasma insulin concentrations to a steady-state and maintained glucose concentrations at/or slightly lower than the individual subjects baseline reading. For each subject two 18G cannulas were inserted, one in the antecubital fossa for insulin and glucose infusions, and one for pharmacokinetic (PK) and blood glucose sampling.
- C-peptide: A euglycaemic/hyperinsulinaemic clamp involves acutely raising the plasma insulin levels to a steady state and maintaining a state of euglycaemia with a glucose infusion, thereby effectively stopping endogenous glucose and insulin production, and as a result reducing the release of C-peptides. This technique will firstly test whether hyperinsulinaemia has an effect on QT interval, and secondly whether C-peptide levels play any role in the proposed effect on the QT interval.
Arm/Group | Insulin Clamp | Glucose | C-peptide
Number analyzed (Participants) | 32 | 32 | 32
msec | -0.01 [-0.02 to 0.04] | -0.86 [-1.45 to -0.27] | -0.71 [-0.98 to -0.45]

5. Secondary Outcome: The QTcF Profile of Oral Moxifloxacin (400 mg) in Healthy Japanese Versus Caucasian Subjects
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4 and 6 hours post-dose
Measure: Mean (95% Confidence Interval); unit: ms
Groups:
- Caucasian Fasted Group: The results of concentration-effect analysis: the effect of moxifloxacin on QTcF (double difference of QTcF) at the time point of maximum mean concentrationof moxifloxacin (1h)
- Caucasian Fed Group; Japanese Fasted Group; Japanese Fed Group: The results of concentration-effect analysis: the effect of moxifloxacin on QTcF (double difference of QTcF) at the time point of maximum mean concentrationof moxifloxacin (4h)
Arm/Group | Caucasian Fasted Group | Caucasian Fed Group | Japanese Fasted Group | Japanese Fed Group
Number analyzed (Participants) | 13 | 13 | 19 | 19
ms | 9.0 [3.2 to 14.7] | 13.7 [8.2 to 19.2] | 17.3 [13.9 to 20.6] | 10.1 [5.1 to 15.1]

ADVERSE EVENTS:
Time Frame: The AEs were recorded at screening: Days: -21 to -3, daily through Period 1 (from Day -2 to Day 3), washout period (3 days), daily through Period 2 (from Day -2 to Day 3) and at follow-up visit (7-14 days after the end of Period 2).
Description: Regular safety assessments have been done by using the following methods: investigator assessment, blood pressure and ECG measurements (12 time points per day in-house), laboratory testing (biochemistry and urinalysis on Day 3 of each period).
Groups:
- Moxifloxacin 400 mg Fasted: Moxifloxacin fasted: One single dose of 400mg moxifloxacin after fasting - This is the standard probe for the assessment of assay sensitivity in Thorough QT (TQT) studies.
  No significant other Adverse Events have been reported.
- Moxifloxacin 400 mg Fed: Moxifloxacin with food: Currently, there is no published data showing the effects of a single 400 mg oral dose of moxifloxacin on the ECG/QT/QTc after food.
  No significant other Adverse Events have been reported.
Arm/Group | Moxifloxacin 400 mg Fasted | Moxifloxacin 400 mg Fed
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
Our findings based on the confirmatory and concentration-effect analysis suggest that any difference between ethnicities was most likely attributable to differences in plasma concentrations and not differences in sensitivity to moxifloxacin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes